CLINICAL TRIAL: NCT02428673
Title: Effects of Standing on Non-Ambulatory Children With Neuromuscular Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gillette Children's Specialty Healthcare (Other)
Responsible Party: Principal Investigator, Walter Truong, Pediatric Orthopedic Surgeon, Gillette Children's Specialty Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Truong POSNA
Record Dates: First submitted 2015-01-07; First posted 2015-04-29 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Osteopenia; Spinal Muscular Atrophy; Cerebral Palsy; Muscular Dystrophy; Spina Bifida; Rett Syndrome
Keywords: Osteopenia; spinal muscular atrophy; cerebral palsy; muscular dystrophy; spina bifida; Rett Syndrome
MeSH Terms: conditions — Bone Diseases, Metabolic; Muscular Atrophy, Spinal; Cerebral Palsy; Muscular Dystrophies; Spinal Dysraphism; Rett Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Load-measuring platform (Other): A load-sensing platform will be placed under each foot of the subject to record the time course of load borne by each of the lower extremities during weight-bearing training in an assisted standing device.
  Interventions: Other: Assisted Standing Treatment Program

INTERVENTIONS:
Other: Assisted Standing Treatment Program

SUMMARY:
Children with neuromuscular disabilities and limited ambulation are at significant risk for decreased bone mineral density (BMD) and increased incidence of fracture. This is caused, in part, by low levels of load experienced by the skeleton due to a child's functional limitations. Low BMD has been shown to be predictive of fracture, and in fact, fractures usually occur without significant trauma in children with neuromuscular conditions. The discomfort and distress from fractures in this population are considerable, and the associated costs to the family and healthcare system are substantial. Numerous interventions have been devoted to improving BMD in these children. Stationary assisted standing devices are widely used and represent the standard-of-care. However, evidence supporting this approach is limited due to inadequate study designs with insufficient numbers of patients.

This study will use load-sensing platforms in patients with neuromuscular conditions. Successful completion of this pilot study will assist in the development of a future multicenter clinical trial to definitively determine relationships, if any, between passive standing and measures of BMD, fracture incidence, pulmonary function, and health-related quality-of-life measures in children with a variety of neuromuscular disabilities (e.g., spinal muscular atrophy, cerebral palsy, muscular dystrophy, spina bifida, Rett syndrome).

Hypothesis: Assisted standing treatment program will gradually increase their duration of standing by up to 75% after the baseline phase.

DETAILED DESCRIPTION:
Children with neuromuscular disabilities and limited ambulation are at significant risk for decreased bone mineral density (BMD) and increased incidence of fracture. This is caused, in part, by low levels of load experienced by the skeleton due to a child's functional limitations. Low BMD has been shown to be predictive of fracture, and in fact, fractures usually occur without significant trauma in children with neuromuscular conditions such as cerebral palsy, spinal muscular atrophy, or other muscular dystrophies. The discomfort and distress from fractures in this population are considerable, and the associated costs to the family and healthcare system are substantial. Numerous interventions have been devoted to improving BMD in these children. Stationary assisted standing devices are widely used and represent the standard-of-care. However, evidence supporting this approach is limited due to inadequate study designs with insufficient numbers of patients.

Various modifications are added to assisted-standing devices to allow children with neuromuscular impairments to achieve standing postures. These customizations lead to load-sharing with the standing device, and consequently, a decrease in the amount of load passing through the lower extremities. Previous investigators developed custom-made load-measuring sensors to quantify the amount of load borne by the lower extremities while in passive standers, and found that the actual load varied from 23-102% of the child's body weight. These load-measuring sensors were specifically developed for restricted laboratory testing, rather than recording the load magnitude and duration of standing in any brand of standing device during daily use at home, school or therapy.

We previously developed load-sensing platforms that accurately measure loads experienced by the lower extremities of children with cerebral palsy in passive standers. These platforms can be incorporated into any stander design, are able to be used on a routine basis at a child's home, school or therapy, and are able to record the duration of weight-bearing to monitor compliance.

This study will use these load-sensing platforms in patients with neuromuscular conditions. Successful completion of this pilot study will assist in the development of a future multicenter clinical trial to definitively determine relationships, if any, between passive standing and measures of BMD, fracture incidence, pulmonary function, and health-related quality-of-life measures in children with a variety of neuromuscular disabilities (e.g., spinal muscular atrophy, cerebral palsy, muscular dystrophy, spina bifida, Rett syndrome).

ELIGIBILITY:
Inclusion Criteria:

1. Must have a neuromuscular condition
2. Must be between 3-14 years old
3. Gross Motor Function Classification System (GMFCS) Level IV or V
4. Must be on a standing treatment program
5. Parent must be able to provide consent

Exclusion Criteria:

1. Currently taking bisphosphonates

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) (measured by DXA) | 10 months
  Change from baseline in BMD, as , at 10 months.
Bone Architecture (measured by pQCT) | 10 months
  Change from baseline in bone architecture, as measured by pQCT, at 10 months.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) | 10 months
  Change from baseline in PedsQL scores at 10 months.
Neuromuscular Module of the PedsQL | 10 months
  Change from baseline in PedsQL neuromuscular module scores at 10 months.
Change in pulmonary function test | 10 months
  Change from baseline in pulmonary function at 10 months.
Change in Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD) | 10 Months
  Change from baseline in CPCHILD score at 10 months.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Truong, MD, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (1):
- Gillette Children's Specialty Healthcare, Saint Paul, Minnesota, United States